CLINICAL TRIAL: NCT02015910
Title: Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy of Januvia (Sitagliptin) in Healing Chronic Diabetic Foot Ulcers
Brief Title: Januvia (Sitagliptin) in Healing Chronic Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by the sponsor due to slow enrollment
Sponsor: Georgetown University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Paul J. Kim, DPM, Doctor of Podiatric Medicine, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISP-RC50959
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Januvia (Sitagliptin) (Experimental): Sitagliptin 100 mg a day for 12 weeks
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Comparison of Sitagliptin a dipeptidyl-peptidase four (DPP-4) inhibitor 100mg pill with placebo comparator
  Other Names: Januvia
  Arms: Januvia (Sitagliptin)
Drug: Placebo — Sugar pill manufactured to mimick Sitagliptin 100mg pill.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to compare the rate of healing as well as percent of wounds healed in Type II diabetic patients with chronic foot ulcerations receiving sitagliptin versus placebo.

The hypothesis for this study is that subjects receiving daily doses of sitagliptin in combination with their regular antihyperglycemic medications will result in increased healing rates as well as a greater number of healed wounds as compared to subjects receiving placebo and their regular antihyperglycemic medications.

DETAILED DESCRIPTION:
Diabetes and diabetes related complications are a major cost burden on the healthcare system encompassing 1/5 of the overall healthcare dollars in the United States [1]. Much of the costs are related to the treatment of lower extremity wounds in the diabetic patient which accounts for 60% of all nontraumatic amputations that are performed [2]. Amputation is often preceded by a chronic ulceration. The incidence of diabetic ulcers is approximately 6% over a 3 year period [1]. Diabetic foot ulcerations are particularly challenging to heal due to a host of factors including vascular compromise, peripheral neuropathy, and begin prone to infection. Therefore, strategies to heal these wounds as quickly as possible are of paramount importance.

Current strategies for chronic wound healing are limited to topical ointments/therapies, allografts/xenografts with or without cell impregnation, dressings, and wound healing devices. None of these current modalities have been shown to be clearly more effective than another [3,4]. Currently, oral medications have not been examined for healing of these chronic ulcerations. Particularly, antihyperglycemic medications have not been studied specifically for the purpose of wound healing. Glucose control and wound healing have been shown to be related [5-7]. However, it is thought that wound healing as a result of tighter glucose control is merely a global effect rather than a direct result of the medications utilized with no evidence that indicates that a specific antihyperglycemic medication works better than another. Further, the mechanism of how and why this relationship exists is not well understood. Specifically, how the microenvironment of the wound as evidenced by changes in the biomarkers has not been delineated.

Januvia (sitagliptin) is an FDA approved antihyperglycemic drug that inhibits the enzyme dipeptidyl peptidase 4 (DPP-4), which is an enzyme that is responsible for the breakdown of glucagon-like peptide (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP). By blocking this effect, GLP-1 and GIP stimulates the secretion of insulin and suppresses the release of glucagon thereby normalizing blood glucose. The unique properties of this drug decrease the likelihood of hypoglycemia. Therefore, this drug is often used in combination of other antihyperglycemic medications to produce a synergistic effect.

DPP4 is expressed on the membranes of a variety of cell types as well as in soluble form, and cleaves the two N-terminal amino acids, X-ala or X-pro, from a limited number of peptide substrates, usually resulting in their inactivation. A family of DPP4 inhibitors, gliptins, have been shown to preserve the full-length active forms of GLP1 and GIP in patients with type II diabetes, enhancing antihyperglycemic activity. In addition to GLP1 and GIP, important substrates of DPP4 essential for wound healing, and altered in diabetes, include SDF-1α/β (stromal cell derived factor 1), PYY (peptide YY), NPY (neuropeptide Y), GM-CSF (granulocyte macrophage colony stimulating factor), G-CSF (granulocyte colony stimulating factor), and IL3 (interleukin 3) [8-12]. SDF, PYY, and NPY are all important for angiogenesis, while GM-CSF, G-CSF, and IL3 are necessary for leukocyte proliferation and infiltration in the wound bed. The observation that DPP4 can cleave and inactive all of these signaling molecules in vivo suggest that modulation of DPP4 activity will have a direct effect on wound healing.

The prospect that a daily oral medication that improves overall glucose control of a diabetic patient as well as expediting the wound healing process is profound. This study explores this possibility.

This is a prospective, randomized study examining the ability of sitagliptin in expediting the wound healing process in the diabetic patient with a chronic foot wound. This is a single center study of 250 total subjects randomized into 2 arms. It is projected that this study will take 3 years to complete. The two arms will be 1) Januvia (sitagliptin) 100mg q day* and 2) placebo-control q day. Patients with Type II diabetes with a chronic foot ulcer will be enrolled into this study. Each subject will be randomized into one of the two arms and will participate in the study for a maximum of 16 weeks. At the end of 16 weeks subjects will be exited from the study. If at any time during the course of the study the wound heals, the subject will be exited from the study after a 2-week confirmatory visit.

*For moderate renal failure subjects, the sitagliptin dose will be adjusted to 50mg q day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age >18
* Type II Diabetes with glycated hemoglobin (hemoglobin A1C) of < 11
* Currently on an oral hyperglycemic medication other than sitagliptin
* A chronic wound defined as the lack of wound healing progress of <15% per week or 50% over a month period
* Ankle brachial index of > 0.80
* Wound located on the foot or ankle (Wagner Grade 1,2)
* Able to comply with the requirements of the research trial

Exclusion Criteria:

* Current use of dipeptidyl-peptidase four (DPP-4) inhibitor or glucagon like peptide one (GLP-1)agonist
* End stage renal disease
* Currently enrolled in another research trial that involves treatment of the wound
* Active infection of the wound
* Wound that probes to bone with osteomyelitis (Wagner Grade 3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Kim, DPM, Principal Investigator — Georgetown University
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data was not collected for use in future research and will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Januvia (Sitagliptin) | Placebo
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Januvia (Sitagliptin) | Placebo | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 68 (0) | 68 (0)
Gender [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Wounds Healed
Description: Compare the rate of healing as well as percent of wounds healed in Type II diabetic patients with chronic foot ulcerations receiving sitagliptin versus placebo.
Time Frame: 12 weeks
Population: Data analysis not completed due to insufficient enrollment.
Arm/Group | Januvia (Sitagliptin) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Januvia (Sitagliptin) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Data was collected for one subject but could not be analyzed due to insufficient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No